CLINICAL TRIAL: NCT04630249
Title: Pilot RCT of Remote Mental Health and Substance Use Screening, Brief Intervention and Referral to Treatment (SBIRT), Compared to In-Person SBIRT for Peripartum Women
Brief Title: Pilot Randomized Controlled Trial (RCT): Remote SBIRT Vs. In-Person SBIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Constance Guille, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00103742
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy; Substance Use; Depression; Anxiety
Keywords: Pregnancy; Depression; Substance Use; Anxiety
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders | interventions — Gravidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Listening to Women and Pregnant and Postpartum People (Experimental): Participants are enrolled in text message-based screenings with immediate automated feedback, paired with remote care coordination and, if appropriate, home-based telemedicine mental health and substance use disorder treatment services. The text screenings contain the SBIRT which is a survey with 9 questions related to depression, anxiety, substance abuse (alcohol, cigarettes, other drugs including prescription medication), and domestic violence.
  Interventions: Behavioral: Listening to Women and Pregnant and Postpartum People
- Usual Care (No Intervention): This group will receive in-person screening and referral to treatment by a nurse or physician per usual prenatal care. The in person screenings contain the SBIRT which is a survey with 9 questions related to depression, anxiety, substance abuse (alcohol, cigarettes, other drugs including prescription medication), and domestic violence.

INTERVENTIONS:
Behavioral: Listening to Women and Pregnant and Postpartum People — Participants are enrolled in text message-based screenings with immediate automated feedback, paired with remote care coordination and, if appropriate, referral to telemedicine mental health and substance use disorder treatment services.
  Arms: Listening to Women and Pregnant and Postpartum People

SUMMARY:
Specific Aim 1: Conduct a pilot, small-scale randomized controlled trial to examine feasibility and preliminary efficacy of LTW, compared to TAU. Outcomes related to feasibility include percentage of eligible patients recruited, study attrition, study retention, and mental health and substance use treatment appointment attendance. Outcomes related to preliminary efficacy will include participation in screening, referral and treatment at baseline, compared to TAU.

Specific Aim 2: Conduct a randomized controlled trial to examine the effectiveness of LTW, compared to TAU. Outcomes related to effectiveness include screening, screening positive, referred to and attendance to treatment at baseline, compared to TAU.

DETAILED DESCRIPTION:
Participants: 450 adult, pregnant or postpartum women

Intervention: Listening to Women is a mobile phone-based program designed to enhance delivery of Screening, Brief Intervention, and Referral to Treatment (SBIRT), an evidence-based approach for mental health and substance use screening and treatment for perinatal women. This program was created as a result of key informant interviews with obstetric providers and pregnant and postpartum women with opioid use disorders. The program utilizes mobile phone text message-based screenings with immediate automated feedback, paired with remote care coordination and, if appropriate, home-based telemedicine mental health and substance use disorder treatment services.

Design: Specific aim 1: A two arm pilot RCT (N=35) with 2:1 allocation will examine feasibility and preliminary efficacy of LTW, compared to TAU. Specific aim 2: A RCT (N=415) with 1:1 allocation will examine effectiveness of LTW, compared to TAU.

This study is part of the HEAL Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

1) age 18-41; 2) currently pregnant or postpartum; 3) if pregnant, receiving prenatal care; 4) English fluency; 5) owner of a cell phone with short message service (SMS) text-message based capability; 6) access to Wireless Fidelity (WIFI) and a device to allow audio and video teleconferencing; 7) able to provide informed consent.

Exclusion Criteria: None

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 415 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Started | 224 | 191
Completed (Follow-up data was extracted from the EHR and may not capture all participants that did not continue prenatal care in the study healthcare system.) | 224 | 191
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care | Total
Number analyzed (Participants) | 224 | 191 | 415
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [27 to 34] | 31 [26 to 34] | 31 [27 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 191 | 415
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 70 | 71 | 141
  Hispanic | 12 | 8 | 20
  Non-Hispanic White | 135 | 110 | 245
  Other | 7 | 2 | 9
Annual Household Income [Count of Participants; unit: Participants]
  Under $25,000 per year | 46 | 31 | 77
  $25,000 per year or more | 178 | 160 | 338
Rurality of Patient's Residence [Count of Participants; unit: Participants]
  Rural | 14 | 18 | 32
  Partially Rural | 154 | 141 | 295
  Urban | 42 | 28 | 70
  Data Missing | 14 | 4 | 18
Number of Living Children [Median (Inter-Quartile Range); unit: children] | 1 [1 to 2] | 1 [0 to 2] | 1 [1 to 2]
Number of Pregnancies [Median (Inter-Quartile Range); unit: pregnancies] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Currently Pregnant [Count of Participants; unit: Participants] | 102 | 85 | 187
Number of Weeks Pregnant [Median (Inter-Quartile Range); unit: weeks] — Population: Pregnant participants only.
  weeks
    number analyzed (Participants) | 102 | 85 | 187
    (all) | 28.0 [20.0 to 33.0] | 28.0 [23.0 to 32.0] | 28.0 [22.0 to 33.0]
Number of Months Postpartum [Median (Inter-Quartile Range); unit: months] — Population: Postpartum participants only.
  months
    number analyzed (Participants) | 122 | 106 | 228
    (all) | 2.0 [1.0 to 4.5] | 2.0 [1.0 to 8.0] | 2.0 [1.0 to 5.0]
Self-Reported Psychiatric Diagnoses [Count of Participants; unit: Participants]
  Mood Disorder | 35 | 27 | 62
  Anxiety Disorder | 67 | 52 | 119
  Substance Use Disorder | 21 | 9 | 30
  Psychotic Disorder | 0 | 0 | 0
  None | 141 | 129 | 270
Self-Reported EPDS Score [Median (Inter-Quartile Range); unit: units on a validated scale] — Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report screening questionnaire where each item is scored from 0 to 3 with a range of possible scores totaling between 0 and 30. The scores measure the severity of postpartum depression. Higher scores indicate greater severity with a total score higher than 10 indicating possible depression.
  units on a validated scale | 5.0 [2.0 to 8.0] | 6.0 [3.0 to 9.0] | 5.0 [3.0 to 9.0]
Self-Reported GAD-7 Score [Median (Inter-Quartile Range); unit: units on a validated scale] — The Generalized Anxiety Disorder scale-7 (GAD-7) is a 7 item diagnostic tool with each item receiving a score between 0 and 3 measure the severity of anxiety symptoms. The total possible range of scores is between 0 and 21 with 0-4 indicating minimal anxiety, 5-9 indicating mild anxiety, 10-14 indicating moderate anxiety and 15-21 indicating severe anxiety.
  units on a validated scale | 3.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 6.0]

OUTCOME MEASURES:

1. Primary Outcome: Completion of SBIRT (Specific Aim 1)
Description: We will compare the proportion of participants that complete a screen for mental health and substance use among those assigned to LTWP, compared to TAU.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 224 | 191
Participants | 221 | 63

2. Primary Outcome: Screened Positive (Specific Aim 1)
Description: We will compare the proportion of those screening positive that are referred to treatment among those assigned to LTWP, compared to TAU.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 224 | 191
Participants | 121 | 11

3. Primary Outcome: Referred to Treatment (Specific Aim 1)
Description: We will compare the proportion of participants referred to treatment that had at least one mental health and/or substance use disorder treatment appointment among those assigned to LTWP, compared to TAU.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 224 | 191
Participants | 31 | 2

4. Primary Outcome: Treatment Attendance (Specific Aim 1)
Description: Treatment attendance (defined as attending at least 1 or more visits with a mental health and/or substance use disorder (SUD) treatment provider during pregnancy and the postpartum year)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 224 | 191
Participants | 20 | 1

5. Secondary Outcome: Screened Positive (Specific Aim 2)
Description: Among those that completed a screen, proportion of participants that screened positive.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 221 | 63
Participants | 121 | 11

6. Secondary Outcome: Referred to Treatment (Specific Aim 2)
Description: Among those that completed a screen, proportion of participants that were referred to treatment.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 221 | 63
Participants | 31 | 2

7. Secondary Outcome: Treatment Attendance (Specific Aim 2)
Description: Among those that completed a screen, proportion of participants that attended a mental health or substance use treatment appointment.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Listening to Women and Pregnant and Postpartum People | Usual Care
Number analyzed (Participants) | 221 | 63
Participants | 20 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the participant's randomization date through 3 months post randomization.
Description: Events related to hospitalization for labor and delivery were not reported as serious adverse events and adverse events.
Groups:
- Treatment as Usual: This group will receive in-person screening and referral to treatment by a nurse or physician per usual prenatal care. The in person screenings contain the SBIRT which is a survey with 9 questions related to depression, anxiety, substance abuse (alcohol, cigarettes, other drugs including prescription medication), and domestic violence.
Arm/Group | Listening to Women and Pregnant and Postpartum People | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/191
Serious Adverse Events (participants affected / at risk) | 3/224 | 3/191
Other Adverse Events (participants affected / at risk) | 0/224 | 0/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Listening to Women and Pregnant and Postpartum People (N=224) | Treatment as Usual (N=191)
Hospitalization etiology unknown (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystectomy (Hepatobiliary disorders) | 3 (3) | 0 (0) — event not related to the intervention
Percutaneous umbilical blood sampling-Intrauterine Transfusion (PUBS-IUT) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Mastitis with Abscess (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limited data capture of primary outcomes in EHR, particularly for treatment attendance. Treatment may have occurred in other settings not captured by EHR. It is possible that participants in TAU were screened and referred but findings were not recorded in the EHR. The study took place within a single health system and findings may not be generalizable. It is unknown whether the screening completion rates within LTWP would differ in settings where staff do not enroll patients into LTWP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT04630249/Prot_001.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04630249/SAP_002.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT04630249/ICF_000.pdf